CLINICAL TRIAL: NCT05449834
Title: Fibrinogen Early In Severe Trauma StudY II
Acronym: FEISTY II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Blood Synergy Program (Unknown); Australian and New Zealand Intensive Care Society Clinical Trials Group (Network); Australasian College for Emergency Medicine (Other); Australian Red Cross Lifeblood (Unknown); Australasian Trauma Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANZIC-RC/ZM001
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Trauma; Haemorrhagic Shock; Coagulopathy
Keywords: Fibrinogen; Cryoprecipitate
MeSH Terms: conditions — Wounds and Injuries; Shock, Hemorrhagic; Hemostatic Disorders | interventions — Fibrinogen; cryoprecipitate coagulum

STUDY DESIGN:
Intervention Model Description: A prospective phase III, multi-centre, randomised, controlled, two arm parallel, open label trial evaluating the effect of FC compared to standard care (Cryo) in severely injured bleeding adult trauma patients with major haemorrhage and hypofibrinogenemia.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: It is not possible to blind the treating clinician to the randomised arm assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibrinogen Concentrate (FC) (Experimental): Fibrinogen Replacement using 3g Fibrinogen Concentrate as per:
  ROTEM FIBTEM A5 ≤ 10mm or TEG FF A10 ≤ 15mm or FibC ≤ 2g/L
  Interventions: Drug: Fibrinogen Concentrate
- Cryoprecipitate (Cryo) (Active Comparator): Fibrinogen Replacement using 10 Units WB or 4U Apheresis Cryo (Australia) as per:
  ROTEM FIBTEM A5 ≤ 10mm or TEG FF A10 ≤ 15mm or FibC ≤ 2g/L
  Interventions: Other: Cryoprecipitate

INTERVENTIONS:
Drug: Fibrinogen Concentrate — 3g Fibrinogen Concentrate
  Other Names: Riastap
  Arms: Fibrinogen Concentrate (FC)
Other: Cryoprecipitate — 10U WB or 4U Apheresis Cryoprecipitate
  Arms: Cryoprecipitate (Cryo)

SUMMARY:
Annually over 7000 Australians are treated for severe trauma. Haemorrhage secondary to severe trauma is a major cause of potentially preventable death and poor outcomes in Australian adults. Severe trauma may trigger changes in blood clotting mechanisms and factor levels leading to inhibition of clot formation and reduced clot strength. This results in the inability of the severely injured trauma patient to form adequate clots to help stop bleeding. There is good evidence to suggest the loss of clotting factors during haemorrhage is associated with worse outcomes and it is thought the early replacement of these factors may reduce bleeding and improve patient outcomes. Fibrinogen is a key clotting factor that helps bind clots together and early fibrinogen replacement may improve outcomes.

Currently fibrinogen is replaced using cryoprecipitate, a blood product made from blood donated by healthy donors which is a precious resource. It can take a significant amount of time to administer as it is frozen and stored in the blood bank. Timely administration of cryoprecipitate is difficult as it requires thawing prior to transfusion. The large doses of cryoprecipitate used in traumatic haemorrhage can put strain on local blood banks in supplying requested units in a timely manner. Additionally, the widely dispersed population of Australia introduces logistic challenges to the maintenance of adequate cryoprecipitate stocks to individual hospital blood banks, especially in remote regions. However, cryoprecipitate contains a number of other coagulation factors (not just fibrinogen) that may be instrumental in clot formation and resistance to fibrinolysis.

Fibrinogen concentrate is an alternative product used to assist in blood clotting. It is a dry powder form of fibrinogen and can be reconstituted at the bedside and given quickly. The use of a fibrinogen factor concentrate with a long shelf life that is easy to use has significant implications for both large urban metropolitan areas and remote isolated communities.

The timing and mode of fibrinogen replacement in traumatic haemorrhage has implications for patient outcomes, blood product availability, costs and the national blood supply. Despite the importance of fibrinogen replacement in traumatic haemorrhage, there have been no clinical trials powered for clinical outcomes directly comparing fibrinogen concentrate and cryoprecipitate. FEISTY II will evaluate the efficacy, safety and cost-effectiveness of Fibrinogen Concentrate vs Cryoprecipitate in trauma patients with major haemorrhage.

FEISTY II is a phase III randomised trial which will enrol 850 patients from Australian and New Zealand major trauma centres, with a primary patient outcome of days alive out of hospital at day 90 after injury. Severely injured trauma patients who require blood transfusion and have evidence of low fibrinogen levels will be randomised to receive either fibrinogen concentrate or standard care with cryoprecipitate

ELIGIBILITY:
Inclusion Criteria:

1. Adult affected by trauma (≥18yrs)
2. Judged to have active haemorrhage by treating clinician
3. Activation of local MHP and/or Transfusion of Emergency Blood Products
4. FIBTEM A5 ≤ 10mm or TEG FF A5 ≤ 15mm or FibC ≤ 2 g/l

Exclusion Criteria:

1. Injury judged incompatible with survival
2. Randomisation unable to occur within 6 hours of presentation to hospital
3. Known pregnancy
4. Known genetic or drug induced coagulation disorder
5. Known objection to blood products
6. Dedicated prior fibrinogen replacement
7. Participation in a competing study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Days Alive and Out of Hospital at 90 Days | 90 Days
  DAOH 90

SECONDARY OUTCOMES:
Number RBC Units at 24 hours | 24 hours
  Red Blood Cells
All cause mortality at 90 days | 90 days
  Mortality at Day 90
All cause mortality at 6 and 24 hours | 24 hours
  Mortality at 6 and 24 hours
Death from haemorrhage at 6 and 24 hours | 24 hours
  Haemorrhage as cause of death at 6 and 24 hours
Ventilator free days up to day 28 | 28 days
  VFD 28 days
Symptomatic thromboembolic events to 28 days | 28 days
  Venous and Arterial Thrombotic events
Quality of life at 3, 6 and 12 months | 12 Months
  EQ5D-5L European Quality of Life 5 Dimensions 5 Levels Scored 0-100, where 0 = Worst QOL and 100 = Best QOL
Health and disability at 3, 6 and 12 months | 12 months
  WHODAS 2.0 World Health Organisation Disability and Assessment Schedule 2.0 Scored 0-100, where 0 = No Disability and 100 = Full Disbility
Functional outcome (Patients with TBI) at 12 months | 12 months
  GOSE Glasgow Outcome Scale Extended Scored 1-8, where 1 = Death and 8 = Upper Good Recovery
Organ failure assessment | 28 days
  Denver MOF Score Denver Multiple Organ Failure Score Scored 0-12, where 0 = No Organ Failure and 12 = Severe MOF

CONTACTS AND LOCATIONS:
Overall Officials: Zoe McQuilten, MBBS, Principal Investigator — Monash University
Locations (24):
- Australia (20):
  - John Hunter Hospital, Newcastle, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Royal Darwin Hospital, Darwin, Northern Territory
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - Sunshine Coast University Hospital, Sunshine Coast, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (4):
  - Aukland City Hospital, Auckland, Aukland
  - Middlemore Hospital, Auckland, Aukland
  - Waikato Hospital, Hamilton, Hamilton
  - Wellington Hospital, Wellington, Wellington Region

IPD SHARING:
Plan to Share IPD: No
No current plan to make IPD available

REFERENCES:
- [Derived] Fatovich DM, Carey S, Iliff J, Jowitt T, Weber DG, Vance JS. Integrating Research Practice Into Resuscitation Simulation Training Improves Recruitment Into Complex Clinical Trials. Emerg Med Australas. 2025 Jun;37(3):e70064. doi: 10.1111/1742-6723.70064. PMID 40420619